CLINICAL TRIAL: NCT01066949
Title: Behavioral Intervention and Adherence in Dialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Alan J. Christensen, Professor, Department of Psychology, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DK72325; R01DK072325 (NIH)
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Kidney Disease
Keywords: hemodialysis; behavior change; patient adherence; self management
MeSH Terms: conditions — Renal Insufficiency, Chronic; Patient Compliance | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Support and discussion (Active Comparator): The Support and Discussion protocol will consist of two integrated components: (a) brief educational materials presented at the start of each session, and (b) group leader facilitated discussion following presentation of the educational materials.
  Interventions: Behavioral: Support and discussion
- Behavioral Self management (Experimental): Self-Regulation group sessions will be generally highly leader-directed though participants will be regularly encouraged to share their experiences dealing with the dialysis regimen. A consistent attempt will be made to focus all group discussion on self-regulatory principles as they relate to treatment adherence.Session material utilized by group-leaders will be highly structured and detailed across the seven sessions.
  Interventions: Behavioral: Behavioral self mangement

INTERVENTIONS:
Behavioral: Behavioral self mangement — Seven weekly, hour long group sessions focused on enhancing patient behavioral self management skills.
  Arms: Behavioral Self management
Behavioral: Support and discussion — Seven, weekly hour long group sessions focused on information provision and supportive discussion amongst participants
  Arms: Support and discussion

SUMMARY:
The aim of the proposed work is to conduct a randomized controlled trial (RCT) evaluation of a behavior change intervention designed to enhance fluid-intake adherence (compliance) among hemodialysis patients. Patient non-adherence (non-compliance) with fluid-intake restrictions is a highly pervasive problem in the hemodialysis population with substantial consequences in terms of increased patient morbidity and mortality. Given the prevalence and clinical importance of adherence among ESRD patients, the design and evaluation of interventions to improve patient adherence is critically important. Surprisingly, however, little such empirical work has been conducted in this area.

The proposed RCT involves testing the efficacy of a behaviorally based, group-administered, "behavioral self regulation" intervention designed to increase adherence to fluid intake restrictions among hemodialysis patients. This structured intervention is designed to be delivered by healthcare providers in a clinical setting to groups of 4-10 patients over seven, one-hour weekly sessions. This study will compare the effect of the structured intervention group with the effect of an educational and support group on fluid-intake adherence in a sample of approximately 200 fluid non-adherent center hemodialysis patients over a 26-week follow-up period. Both clinical (interdialysis session weight gain) and self-report indices of fluid-intake adherence will be examined. We believe that the proposed research is of potentially very high impact given the high prevalence and clear clinical consequences of hemodialysis patient nonadherence and the potential for a relatively low-cost, structured intervention to significantly reduce this type of maladaptive patient behavior in the hemodialysis treatment context.

DETAILED DESCRIPTION:
Upon consent and enrollment into the study, patients will be given a packet of questionnaires to take home, complete, and return using a postage-paid envelope. These questionnaires will include a patient background form, which includes information on age, gender, marital status, years of education, employment status, and race/ethnicity, and two measure of health beliefs and attitudes (the Krantz Health Opinion Survey and the Multidimensional Health Locus of Control Scale. A copy of all measures in attached to this application.

Following consent and randomization participants will be assigned to one of two comparison study arms. Both study arms involve participation in a weekly, hour-long, patient support group for seven weeks. As described below the groups differ in terms of the content focus.

Patients randomly assigned to the Self-Regulation arm will meet in groups of 4-10 participants at their usual hemodialysis clinic for hour-long weekly sessions for seven weeks. Two to four groups will be conducted at each participating center depending on center size. Groups will be led by a member of the UIHC research team with at least two years previous professional experience with behavior change techniques, at least two years previous experience with the hemodialysis population, and a master's or doctoral level degree in psychology. Each UIHC team group leader will be responsible for 3-4 groups over the duration of the project. Session material utilized by group-leaders will be highly structured and detailed across the seven sessions. Self-Regulation group sessions will be generally highly leader-directed though participants will be regularly encouraged to share their experiences dealing with the dialysis regimen. A consistent attempt will be made to focus all group discussion on self-regulatory principles as they related to treatment adherence. An outline of topics for the Self-Regulation groups is attached.

Patients randomly assigned to the Support and Discussion arm will also meet in groups of 4-10 participants at their usual hemodialysis clinic for hour-long weekly sessions for seven weeks. Two to four groups will be conducted at each participating center depending on center size. These groups will be also led by a member of the UIHC research team, with each group leader responsible for 3-4 groups over the duration of the project. The Support and Discussion protocol will consist of two integrated components: (a) brief educational materials presented at the start of each session, and (b) group leader facilitated discussion following presentation of the educational materials. An outline of topics for the Support and Discussionn groups is also attached.

Patient adherence to the fluid-intake regimen will be determined by computing the amount of weight a patient gained between dialysis treatment sessions (termed "interdialytic weight gain" or IWG) as recorded in the patient's regular medical record. Mean IWG averaged over two weeks (six sessions) at each assessment point will serve as the primary dependent measure in this study. The pre-enrollment assessment (Time 0) will comprise the two weeks immediately preceding the start of group meetings, Time 1 will comprise the two weeks immediately following the final intervention session, Time 2 will comprise the 12th and 13th post-intervention weeks and the Time 3 assessment will consist of the 25th and 26th post-intervention weeks. Patients will also be asked to complete a previously validated self-report assessment of hemodialysis patient adherence to fluid restrictions (Dialysis Diet and Fluid Non-Adherence Questionnaire). This measure assesses fluid-intake adherence over the previous two weeks and will be obtained on a schedule which parallels the collection of the clinical IWG data.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be deemed eligible if they have a mean (averaged over the preceeding four weeks) pre-enrollment, interdialysis weight gain (IWG) greater than 2.5 kg. Other inclusion criteria will include having been receiving hemodialysis for a minimum of three months, patient age over 18 years, and English speaking.

Exclusion Criteria:

* Patients residing in a nursing home/long-term care facility will be excluded from participation primarily due to likelihood of diminished patient self-management of diet and fluid intake in this setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2006-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Interdialysis weight gain | from enrollment to 6 months post-enrollment

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Tri-State Dialysis, Dubuque, Iowa
  - University of Iowa renal dialysis program, Iowa City, Iowa

REFERENCES:
- [Derived] Howren MB, Cozad AJ, Christensen AJ. The interactive effects of patient control beliefs on adherence to fluid-intake restrictions in hemodialysis: Results from a randomized controlled trial. J Health Psychol. 2017 Nov;22(13):1642-1651. doi: 10.1177/1359105316631813. Epub 2016 Feb 22. PMID 26908586
- [Derived] Howren MB, Kellerman QD, Hillis SL, Cvengros J, Lawton W, Christensen AJ. Effect of a Behavioral Self-Regulation Intervention on Patient Adherence to Fluid-Intake Restrictions in Hemodialysis: a Randomized Controlled Trial. Ann Behav Med. 2016 Apr;50(2):167-76. doi: 10.1007/s12160-015-9741-0. PMID 26631085